CLINICAL TRIAL: NCT03531892
Title: Phase III Study of AJM300 in Patients With Active Ulcerative Colitis
Brief Title: A Study to Evaluate the Safety and Efficacy of AJM300 in Participants With Active Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EA Pharma Co., Ltd. (Industry)
Collaborators: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AJM300/CT3; JapicCTI-183924 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2018-05-09; First posted 2018-05-22 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-04

CONDITIONS: Colitis, Ulcerative
Keywords: Ulcerative Colitis; Inflammatory Bowel Disease, Ulcerative Colitis Type; Colitis; AJM300
MeSH Terms: conditions — Colitis, Ulcerative; Colitis | interventions — AJM300

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AJM300 960mg/dose (Experimental): Participants will orally receive AJM300 960 mg tablets, three times daily after meals for 8 weeks.
  Interventions: Drug: AJM300
- Placebo (Placebo Comparator): Participants will orally receive AJM300 placebo-matching tablets, three times daily after meals for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AJM300 — AJM300 film-coated tablets.
  Other Names: Carotegrast methyl
  Arms: AJM300 960mg/dose
Drug: Placebo — Placebo matched to AJM300 tablets.
  Arms: Placebo

SUMMARY:
The study will investigate the efficacy and safety of an oral dose of AJM300 960 milligram (mg)/dose administered three times daily for 8 weeks in participants with active ulcerative colitis.

ELIGIBILITY:
Major Inclusion Criteria:

1. Participants diagnosed with ulcerative colitis.
2. Participants with moderate ulcerative colitis who satisfy all of the following criteria at Day of enrollment.

   1. Mayo Clinic scores of 6-10 .
   2. Endoscopic subscore greater than or equal to (>=) 2.
   3. Rectal bleeding subscore >=1.
3. Participants with inadequate response or intolerant to oral 5-ASA
4. Participants who are capable of providing written informed consent

Major Exclusion Criteria:

1. Participants with extensive detachment of mucosa or deep ulcer.
2. Participants with oral corticosteroid dependency.
3. Participants with a complication of marked reduction of immune function.
4. Participants who were clinically suspected to have a complication of infectious enteritis.
5. Participants with a history or complication of serious infection within 1 year prior to the day of enrollment.
6. Participants with central nervous system (CNS) neurological symptoms.
7. Participants with the following criteria:

   * Serious heart disease
   * Renal impairment
   * Hepatic impairment
8. Participants with a history of serious drug induced allergy with unknown cause.
9. Participants with malignant tumor or those whose treatments were completed in less than 5 years.
10. Participants with apparent psychological signs.
11. Pregnant women, nursing women, women with suspected pregnancy, women who wish to become pregnant during the period from informed consent through to the end of observation/examination at Week 8, and women who do not consent to the use of appropriate birth control methods.
12. Participants who are definitely eligible for surgical intervention such as large bowel perforation, major bleeding, and toxic megacolon syndrome, etc.
13. Participants who are participants of another clinical study including follow-up observation at the time of informed consent.
14. Participants who received another investigational drug within 12 weeks prior to the examinations/observation defined by the protocol.
15. Participants who received investigational drugs in the study of AJM300.
16. Participants determined to be ineligible for participation in this study by the investigator or sub-investigator.

Ages: 16 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Clinical Response Rate Based on Mayo Score | At Week 8
  Clinical response rate is defined by the percentage of participants who satisfy the combined definition of the change of the total value of Mayo score and the change or the actual value of individual subscales. Mayo score is used in clinical trials to assess ulcerative colitis (UC) disease activity. It consists of 4 subscales: stool frequency, rectal bleeding, findings on endoscopy and physician's global assessment. Each subscale is scored on a scale of 0 to 3, where 0= normal condition and 3= severe disease condition. The total Mayo score ranges from 0 to 12, with higher scores indicating more severe disease.

SECONDARY OUTCOMES:
Clinical Remission Rate Based on Mayo Score | At Week 8
  Clinical remission rate is defined by the percentage of participants with Mayo score <=2 and no subscore greater than (>) 1.
Mucosal Healing Rate | At Week 8
  Mucosal healing rate is defined by the percentage of participants with Mayo endoscopic subscore <=1.
Complete Mucosal Healing Rate | At Week 8
  Complete mucosal healing rate is defined by the percentage of participants with Mayo endoscopic subscore =0.
Clinical Response Rate Based on Partial Mayo Score | At Week 8
  Clinical response rate is defined by the percentage of participants who satisfy the combined definition of the change of the total value of partial Mayo score and the change or the actual value of individual subscales. Partial Mayo score is used in clinical trials to assess UC disease activity. It consists of 3 subscales: stool frequency, rectal bleeding and physician's global assessment. Each subscale is scored on a scale of 0 to 3, where 0= normal condition and 3= severe disease condition. The total partial Mayo score ranges from 0 to 9, with higher scores indicating more severe disease.
Clinical Remission Rate Based on Partial Mayo Score | At Week 8
  Clinical remission rate is defined by the percentage of participants with partial Mayo score <=2 and no subscore >1.
Modified Clinical Remission Rate 1 | At Week 8
  Modified Clinical remission rate 1 is defined by percentage of participants who satisfies the three conditions such as: rectal bleeding subscore =0, Stool frequency subscore =0 and Endoscopic subscore <=1.
Modified Clinical Remission Rate 2 | At Week 8
  Modified Clinical remission rate 2 is defined by the percentage of participants who satisfies the three conditions such as: rectal bleeding subscore =0, a decrease in the stool frequency subscore of at least 1 point or an absolute stool frequency subscore of 0 or 1 and Endoscopic subscore <=1.
Percentage of Rectal Bleeding Subscore of 0 | At Week 8
  Percentage of rectal bleeding subscore of 0 means the percentage of participants with rectal bleeding score =0.
Change From Baseline in Mayo score | Baseline, Week 8
  Mayo score is used in clinical trials to assess UC disease activity. It consists of 4 subscales: stool frequency, rectal bleeding, findings on endoscopy and physician's global assessment. Each subscale is scored on a scale of 0 to 3, where 0= normal condition and 3= severe disease condition. The total Mayo score ranges from 0 to 12, with higher scores indicating more severe disease.
Change From Baseline in Partial Mayo Score | Baseline, Week 8
  Partial Mayo score is used in clinical trials to assess UC disease activity. It consists of 3 subscales: stool frequency, rectal bleeding and physician's global assessment. Each subscale is scored on a scale of 0 to 3, where 0= normal condition and 3= severe disease condition. The total Mayo score ranges from 0 to 9, with higher scores indicating more severe disease.
Change From Baseline in Fecal Calprotectin | Baseline, Week 8
Change From Baseline in Peripheral Blood White Blood Cell (WBC) Differentiation (Neutrophil, Eosinophil, Basophil, Lymphocyte, and Monocyte Counts) | Baseline, Week 8

CONTACTS AND LOCATIONS:
Locations (82):
- Japan (82):
  - AJM300/CT3 trial site 41, Nagoya, Aichi-ken
  - AJM300/CT3 trial site 57, Nagoya, Aichi-ken
  - AJM300/CT3 trial site 63, Nagoya, Aichi-ken
  - AJM300/CT3 trial site 9, Toyoake, Aichi-ken
  - AJM300/CT3 trial site 33, Toyohashi, Aichi-ken
  - AJM300/CT3 trial site 42, Toyota, Aichi-ken
  - AJM300/CT3 trial site 39, Hirosaki, Aomori
  - AJM300/CT3 trial site 49, Hirosaki, Aomori
  - AJM300/CT3 trial site 11, Kashiwa, Chiba
  - AJM300/CT3 trial site 51, Kashiwa, Chiba
  - AJM300/CT3 trial site 73, Sakura, Chiba
  - AJM300/CT3 trial site 54, Urayasu, Chiba
  - AJM300/CT3 trial site 81, Matsuyama, Ehime
  - AJM300/CT3 trial site 53, Kurume, Fukuoka
  - AJM300/CT3 trial site 24, Tikushino, Fukuoka
  - AJM300/CT3 trial site 55, Isesaki, Gunma
  - AJM300/CT3 trial site 35, Fukuyama, Hiroshima
  - AJM300/CT3 trial site 18, Asahikawa, Hokkaido
  - AJM300/CT3 trial site 26, Asahikawa, Hokkaido
  - AJM300/CT3 trial site 2, Sapporo, Hokkaido
  - AJM300/CT3 trial site 3, Sapporo, Hokkaido
  - AJM300/CT3 trial site 4, Sapporo, Hokkaido
  - AJM300/CT3 trial site 79, Akashi, Hyōgo
  - AJM300/CT3 trial site 34, Kobe, Hyōgo
  - AJM300/CT3 trial site 64, Nishinomiya, Hyōgo
  - AJM300/CT3 trial site 82, Kasama, Ibaraki
  - AJM300/CT3 trial site 75, Tsukuba, Ibaraki
  - AJM300/CT3 trial site 19, Morioka, Iwate
  - AJM300/CT3 trial site 16, Takamatsu, Kagawa-ken
  - AJM300/CT3 trial site 12, Kamakura, Kanagawa
  - AJM300/CT3 trial site 14, Sagamihara, Kanagawa
  - AJM300/CT3 trial site 32, Sagamihara, Kanagawa
  - AJM300/CT3 trial site 13, Yokohama, Kanagawa
  - AJM300/CT3 trial site 6, Yokohama, Kanagawa
  - AJM300/CT3 trial site 47, Tsu, Mie-ken
  - AJM300/CT3 trial site 46, Yokkaichi, Mie-ken
  - AJM300/CT3 trial site 45, Sendai, Miyagi
  - AJM300/CT3 trial site 50, Sendai, Miyagi
  - AJM300/CT3 trial site 78, Sendai, Miyagi
  - AJM300/CT3 trial site 22, Nagaoka, Niigata
  - AJM300/CT3 trial site 15, Kurashiki, Okayama-ken
  - AJM300/CT3 trial site 70, Kurashiki, Okayama-ken
  - AJM300/CT3 trial site 77, Higashiosaka, Osaka
  - AJM300/CT3 trial site 76, Sayama, Osaka
  - AJM300/CT3 trial site 10, Takatsuki, Osaka
  - AJM300/CT3 trial site 40, Ageo, Saitama
  - AJM300/CT3 trial site 5, Ageo, Saitama
  - AJM300/CT3 trial site 72, Tokorozawa, Saitama
  - AJM300/CT3 trial site 17, Hamamatsu, Shizuoka
  - AJM300/CT3 trial site 60, Ashikaga, Tochigi
  - AJM300/CT3 trial site 29, Shimotsuga, Tochigi
  - AJM300/CT3 trial site 71, Utsunomiya, Tochigi
  - AJM300/CT3 trial site 61, Bunkyo, Tokyo
  - AJM300/CT3 trial site 68, Bunkyo, Tokyo
  - AJM300/CT3 trial site 59, Chiyoda City, Tokyo
  - AJM300/CT3 trial site 30, Chūō, Tokyo
  - AJM300/CT3 trial site 31, Hachiōji, Tokyo
  - AJM300/CT3 trial site 56, Minato, Tokyo
  - AJM300/CT3 trial site 66, Minato, Tokyo
  - AJM300/CT3 trial site 80, Mitaka, Tokyo
  - AJM300/CT3 trial site 38, Shinagawa, Tokyo
  - AJM300/CT3 trial site 21, Shinjuku, Tokyo
  - AJM300/CT3 trial site 52, Shinjuku, Tokyo
  - AJM300/CT3 trial site 8, Shūnan, Yamaguchi
  - AJM300/CT3 trial site 23, Kofu, Yamanashi
  - AJM300/CT3 trial site 44, Chiba
  - AJM300/CT3 trial site 43, Fukuoka
  - AJM300/CT3 trial site 58, Fukuoka
  - AJM300/CT3 trial site 69, Fukuoka
  - AJM300/CT3 trial site 67, Gifu
  - AJM300/CT3 trial site 28, Hiroshima
  - AJM300/CT3 trial site 36, Hiroshima
  - AJM300/CT3 trial site 74, Hiroshima
  - AJM300/CT3 trial site 62, Kyoto
  - AJM300/CT3 trial site 7, Kyoto
  - AJM300/CT3 trial site 48, Nagasaki
  - AJM300/CT3 trial site 65, Okayama
  - AJM300/CT3 trial site 1, Osaka
  - AJM300/CT3 trial site 37, Ōita
  - AJM300/CT3 trial site 20, Saga
  - AJM300/CT3 trial site 25, Saga
  - AJM300/CT3 trial site 27, Toyama

REFERENCES:
- [Derived] Matsuoka K, Watanabe M, Ohmori T, Nakajima K, Ishida T, Ishiguro Y, Kanke K, Kobayashi K, Hirai F, Watanabe K, Mizusawa H, Kishida S, Miura Y, Ohta A, Kajioka T, Hibi T; AJM300 Study Group. AJM300 (carotegrast methyl), an oral antagonist of alpha4-integrin, as induction therapy for patients with moderately active ulcerative colitis: a multicentre, randomised, double-blind, placebo-controlled, phase 3 study. Lancet Gastroenterol Hepatol. 2022 Jul;7(7):648-657. doi: 10.1016/S2468-1253(22)00022-X. Epub 2022 Mar 30. PMID 35366419